CLINICAL TRIAL: NCT07327398
Title: A Randomized, Double-blind, Active-controlled Phase Ⅱ Clinical Trial to Evaluate the Immunogenicity and Safety of the Influenza Virus Split Vaccine for Individuals Aged 60 Years and Above
Brief Title: Phase Ⅱ Clinical Trial of Influenza Virus Split Vaccine for Individuals Aged 60 Years and Above
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-V05-002
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Influenza
Keywords: Influenza virus split vaccine; Safety; Immunogenicity; The elderly
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Influenza virus split vaccine (0.7mL/vial) (Experimental): Influenza virus split vaccine (0.7mL/vial)
  Interventions: Biological: Influenza virus split vaccine (0.7mL/vial)
- Influenza virus split vaccine (Active Comparator): Influenza virus split vaccine
  Interventions: Biological: Influenza virus split vaccine

INTERVENTIONS:
Biological: Influenza virus split vaccine (0.7mL/vial) — Influenza virus split vaccine, with a specification of 0.7mL/bottle, containing 60 μ g of hemagglutinin from H1N1, H3N2, and B influenza virus strains each Control: Influenza virus split vaccine.
  Arms: Influenza virus split vaccine (0.7mL/vial)
Biological: Influenza virus split vaccine — Influenza virus split vaccine, with a specification of 0.5mL/bottle, containing 15 μ g of hemagglutinin from H1N1, H3N2, and B influenza virus strains each.
  Arms: Influenza virus split vaccine

SUMMARY:
To evaluate the immunogenicity of administering one dose of influenza virus split vaccine (0.7mL/dose) to individuals aged 60 and above.

DETAILED DESCRIPTION:
This is a randomized, blinded, parallel controlled trial design, a total of 1200 participants aged ≥ 60 years were enrolled in the study. Study participants were randomly vaccinated with either the experimental vaccine: influenza virus split vaccine (0.7mL/dose) or the control vaccine: influenza virus split vaccine, at a 1:1 ratio. One dose of the vaccine was administered on day 0 for immunogenicity and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old, gender not limited, and able to provide legal identification;
* Volunteers voluntarily participate in the study and sign an informed consent form;
* Volunteers have the ability to understand research procedures, use thermometers, scales, and fill out diary cards as required, and can participate in all planned follow-up visits.

Exclusion Criteria:

* On the day of enrollment, the axillary temperature was ≥ 37.3 ℃;
* Those who have had influenza in the past 6 months or meet the definition of influenza like cases;
* Have received any influenza vaccine within the past 12 months or have planned to receive any influenza vaccine during the study period;
* Allergies to any components of the research vaccine, history of allergic reactions to the use of gentamicin sulfate, history of severe allergies to any vaccine/drug, or history of asthma;
* Suffering from a serious illness that prevents the completion of the entire study; Within 3 days prior to vaccination, there is an acute illness or an acute exacerbation of a chronic disease;
* Have used antipyretic or analgesic drugs or anti allergic drugs within 3 days before vaccination;
* Have received any vaccine within 2 weeks prior to vaccination;
* Have received immunosuppressive therapy or other immunomodulatory drugs within 6 months prior to receiving the experimental vaccine, For example, immunosuppressive doses of glucocorticoids, monoclonal antibodies, thymosin, interferon, etc., or planned to receive such treatment within one month after the first dose of vaccination to full immunization, but local medication is allowed;
* Suffering from congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, or other autoimmune diseases;
* Suffering from serious chronic diseases, serious cardiovascular diseases, such as hypertension that cannot be controlled by drugs, diabetes that cannot be controlled by drugs or has serious complications, liver and kidney diseases, pulmonary edema, malignant tumors, etc;
* Have received blood or blood related products within the past 6 months;
* Individuals with progressive neurological disorders, including a history of seizures, epilepsy, encephalopathy, Guillain Barr é syndrome, psychiatric or family history;
* Have a history of abnormal coagulation function and have been using anticoagulants within 3 weeks before vaccination;
* Patients with splenectomy, functional splenectomy, splenectomy, or other important organ resection or partial resection;
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit;
* Currently or recently planning to participate in other clinical trials;
* Researchers determine any situation that is not suitable for clinical trials.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, the HI antibody seroconversion rate against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.
Ratio of ≥1:40 | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, the ratio of HI antibody titers ≥ 1:40 against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.
Geometric mean titer (GMT) | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, GMT of HI antibodies against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.
Geometric mean increase (GMI) | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, GMI of HI antibodies against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.

SECONDARY OUTCOMES:
Solicited Adverse Events (AEs) | 7 days after vaccination
  Adverse events defined by the protocol that occurred to the participant during 0-7 days after vaccination.
Unsolicited Adverse Events | 30 days after vaccination
  Other adverse events that occurred among participants within 0-30 days after vaccination, in addition to the solicited adverse events.
Serious Adverse Events (SAEs) | 6 months after vaccination
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Danjiangkou City Center for Disease Control and Prevention, Wuhan, Hubei
  - Yunxi County Center for Disease Control and Prevention, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No